CLINICAL TRIAL: NCT01574079
Title: Effect of Mirror Therapy on Lower Extremity Motor Control and Gait in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Lisa J Barnes, Associate Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-0244
Record Dates: First submitted 2012-01-30; First posted 2012-04-10 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): The control group will receive traditional physical therapy interventions directed at neuromuscular rehabilitation.
  Interventions: Other: Traditional Physical Therapy
- Physical Therapy plus Mirror Therapy (Experimental): The mirror therapy will entail 15 minutes of exercises for the lower extremities focusing on ankle dorsiflexion, knee flexion, and hip flexion.
  Interventions: Other: Physical Therapy plus Mirror Therapy

INTERVENTIONS:
Other: Traditional Physical Therapy — Traditional physical therapy includes, but is not limited to, therapeutic exercise, functional mobility training, pre-gait and gait activities, electrotherapeutic modalities, and education.
  Arms: Traditional Physical Therapy
Other: Physical Therapy plus Mirror Therapy — The treatment group will receive traditional physical therapy intervention as described in the control group with the addition of mirror therapy. The participant will attempt to perform the flexion exercises with both lower extremities. The patient will be blinded to the affected lower extremity with a mirror, and will be looking at the image of the unaffected lower extremity superimposed on the affected lower extremity as he or she performs the activities.
  Arms: Physical Therapy plus Mirror Therapy

SUMMARY:
Mirror therapy may be an effective intervention in increasing motor control and gait performance in patients with stroke.

DETAILED DESCRIPTION:
Using a mirrored image of the uninvolved extremity superimposed upon the involved extremity during exercise may facilitate improved motor control in patients after stroke.

ELIGIBILITY:
Inclusion Criteria:

* lower extremity Brunnstrom stage 2,
* lower extremity modified ashworth < 3,
* has the ability to follow 3-step command in English,
* has only unilateral involvement.

Exclusion Criteria:

* lower extremity Brunnstrom stage 1,
* lower extremity modified ashworth 3 or higher,
* history of prior stroke,
* Passive Range of Motion limitation of hip and or knee flexion < 90,
* has visual deficits which prevent participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Barnes, PT DPT, Principal Investigator — University of Mississippi Medical Center; Keri H McCullough, DPT, Study Director — University of Mississippi Medical Center - University Rehabilitation; Kim C Wilcox, PT MsPT PhD, Study Director — University of Mississippi Medical Center - Director of Neurologic Residency Program
Locations (1):
- University of Mississippi Medical Center - University Rehabilitation, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Physical Therapy: The control group will receive traditional physical therapy which includes, but is not limited to, therapeutic exercise, functional mobility training, pre-gait and gait activities, electrotherapeutic modalities, and education.
- Physical Therapy Plus Mirror Therapy: The treatment group will receive traditional physical therapy with the addition of 15 minutes of mirror therapy consisting of lower extremity ankle dorsiflexion, knee flexion, and hip flexion. The participant will attempt to perform the exercises with both lower extremities. The patient will be blinded to the affected lower extremity with a mirror, and will be looking at the image of the unaffected lower extremity superimposed on the affected lower extremity as he or she performs the activities.
Period: Overall Study
Arm/Group | Traditional Physical Therapy | Physical Therapy Plus Mirror Therapy
Started | 18 | 15
Completed | 17 | 13
Not Completed | 1 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Traditional Physical Therapy: The control group received traditional physical therapy which included, but was not limited to, therapeutic exercise, functional mobility training, pre-gait and gait activities, electrotherapeutic modalities, and education.
- Physical Therapy Plus Mirror Therapy: The treatment group received traditional physical therapy with the addition of mirror therapy. The mirror therapy consisted of 15 minutes of exercises for the lower extremities focusing on ankle dorsiflexion, knee flexion, and hip flexion. The participant attempted to perform the exercises with both lower extremities. The participant was blinded to the affected lower extremity with a mirror, and was looking at the image of the unaffected lower extremity superimposed on the affected lower extremity as he or she performed the activities.
- Total: Total of all reporting groups
Arm/Group | Traditional Physical Therapy | Physical Therapy Plus Mirror Therapy | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.47 (11.94) | 48.85 (15.53) | 51.47 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Functional Independence Measure - Locomotor Score
Description: The Functional Independence Measure (FIM)assesses level of disability and measures progress toward independence with rehabilitational intervention. The tool consists of 18 items. Only the the locomotor score was used to assess gait ability in this study. The locomotor score ranges from 1 - 7 with a higher score indicating a higher level of functional independence.
Time Frame: measured at admission and discharge from rehab estimated length of stay 14 days
Population: Thirty-three participants enrolled in the study with 3 dropping out before completion. Two of these were due to medical issues, and one was discharged unexpectedly
Measure: Mean (Standard Deviation); unit: outcome score
Groups:
- Control Group: The control group received traditional physical therapy which included, but was not limited to, therapeutic exercise, functional mobility training, pre-gait and gait activities, electrotherapeutic modalities, and education.
- Treatment Group: The treatment group received traditional physical therapy with the addition of mirror therapy. The mirror therapy consisted of 15 minutes of exercises for the lower extremities focusing on ankle dorsiflexion, knee flexion, and hip flexion. The participant attempted to perform the exercises with both lower extremities. The participant was blinded to the affected lower extremity with a mirror, and was looking at the image of the unaffected lower extremity superimposed on the affected lower extremity as he or she performed the activities.
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 17 | 13
outcome score
  FIM locomotor score on admission | 1.65 (1.06) | 1.33 (0.65)
  FIM locomotor score at discharge | 3.82 (1.38) | 4.25 (0.62)

2. Secondary Outcome: Timed Up and Go
Description: The Timed Up and Go (TUG) is used to assess balance and gait, and to estimate fall risks in patients with deficits. The participant rises from a seated position in a chair, walks 3 meters, turns around, returns to the chair, and sits down. The test is measured in seconds, with a lower number indicating a higher level of independence and the least risk for falls.
Time Frame: Measured at admission and discharge with estimated length of stay 14 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 17 | 13
seconds
  TUG on admission (in seconds) | 100.69 (53.42) | 97.75 (47.69)
  TUG at discharge (in seconds) | 50.6 (34.88) | 49.25 (15.96)

3. Secondary Outcome: Stroke Rehabilitation Assessment of Movement
Description: The Stroke Rehabilitation Assessment of Movement (STREAM)is designed to measure mobility and motor ability after stroke. There are three subscales with 10 items each assessing the upper extremity, lower extremity, and basic mobility. Only the lower extremity and basic mobility items were used in this study. The lower extremity scores ranged from 0 - 18 with higher scores indicating a higher level of motor control. The basic mobility scores ranged from 0 - 30 with high numbers indicating a higher level of functional mobility.
Time Frame: measured at admission and discharge with estimated length of stay 14 days
Measure: Mean (Standard Deviation); unit: outcome score
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 17 | 13
outcome score
  STREAM LE admission | 8.18 (4.97) | 5.33 (1.92)
  STREAM LE discharge | 12.41 (5.33) | 8.58 (2.61)
  STREAM mobility on admission | 6.29 (7.65) | 5.92 (4.42)
  STREAM mobility at discharge | 16.47 (9.86) | 14.67 (6.02)

ADVERSE EVENTS:
Arm/Group | Control Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes